CLINICAL TRIAL: NCT05323331
Title: Effects of Circuit Training Program on Cardiopulmonary Parameters and Functional Capacity in Post COVID 19 Patients
Brief Title: Circuit Training Program in Post COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Hira Haumayun
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Cardiorespiratory Fitness; Functional Fitness; COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit Training (Experimental): This group preformed interval training alternating between aerobic and resistance training, varying between moderate to high intensity. Each set started with 3 minutes of aerobic training on cycle or treadmill followed by resistance training and a rest interval. Eight circuits were formed; horizontal rowing, chest press, leg press, shoulder press, leg extension, lateral pull down, leg flexion and partial squat. Weight was calculated through 1 RM calculation.
  This training is to be carried out for 12 weeks, in three phases, the intensity progressing from light to moderate (30% of RM to 50%). Sessions will be carried out thrice a week.
  Interventions: Other: Circuit Training Exercise Program
- Aerobic Training (Active Comparator): The control group consists of aerobic exercise training, with 20 minutes on the cycle, 15 minutes of treadmill and 10 minutes of walking
  Interventions: Other: Aerobic Training Exercise Program

INTERVENTIONS:
Other: Circuit Training Exercise Program — The participants allocated to this group will perform Circuit Training Exercise Program
  Arms: Circuit Training
Other: Aerobic Training Exercise Program — The participants allocated to this group will perform Circuit Training Exercise Program
  Arms: Aerobic Training

SUMMARY:
The objective of this study will be to compare the effects of Circuit Training Program on Cardiopulmonary Parameters and Functional Capacity in Post COVID 19 patients. This study will be a Randomized Clinical trial. Data will be collected from Boston Physiotherapy and Wellness Clinic, Lahore. One group will receive Circuit Training and other group will receive Aerobic Exercises. All subjects will receive a total of three treatment sessions per week over the period of 12 weeks. Outcome will be measured at baseline, 6th week and 12th week with 6 Minute Walk Test (6MWT), Rate of Perceived Exertion (RPE 6-20), Spirometer for PFT and Post-Covid 10 Functional Status Scale.The data will be analyse using SPSS v 25.

DETAILED DESCRIPTION:
Coronavirus disease (Covid19) caused by SARs Cov-2 is primarily a respiratory condition but it also has many extrapulmonary manifestations leading to persistent symptoms of fatigue, weakness, reduced functional status, aerobic capacity and strength. Patients with cardiovascular and pulmonary comorbidities have varying severity of disease and increased risk of mortality and morbidity. Cardiopulmonary Rehabilitation has been shown to improve the functional capacity and quality of life of patients with cardiac dysfunction and chronic pulmonary conditions in acute, sub-acute and chronic stages of disease. Different modes of exercises including aerobic, resistance, combined aerobic and resistance programs known as circuit training at varying frequencies, intensities and doses are given to these patients according to their symptoms.

Circuit Training program consists of both aerobic and resistance exercises hence it ensures both endurance and strength training during the exercise session. Some researchers have shown that circuit-based resistance training, where lighter loads are lifted with minimal rest, is very effective for increasing maximum oxygen consumption, maximum pulmonary ventilation, functional capacity, and strength while improving body composition Thus, circuit training is a time-efficient training modality that can elicit demonstrable improvements in health and physical fitness.Combined aerobic and resistance training improves peak VO2, muscle strength and HRQoL and should be considered as a component of care of patients of heart failure. The combination of resistance and aerobic modalities has been shown to be the best form of training for individuals with pulmonary conditions like COPD as well as being recommended by international guidelines for the clinical treatment of these patients in rehabilitation programs.

The same principles apply to management of Covid19 patients with inpatient rehabilitation given to acute cases while increasing evidence shows that rehabilitation post-recovery is beneficial to promote early return to function. These studies focus mostly either on aerobic training or resistance exercises; hence this study is aimed towards studying the effects of Circuit Training in post Covid19 population to improve the functional parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Middle age adults (40-60 years), medically stable, but previously diagnosed with cardiac diseases.
2. Patients who have recovered recently from Covid-19 (6-8 weeks post-discharge).
3. Oxygen saturation levels are maintained above 92% at rest and during exercise.
4. Heart Rate should not be elevated more than 20 beats per minute as per the calculated heart rate range (if the patient is on beta-blockers, that should be kept in consideration)
5. Systolic blood pressure should be ≥90 mmHg and ≤180 mmHg.
6. Symptoms of dyspnea: Borg scale >4
7. Fatigue: Rate of Perceived Exertion (RPE) >11-12

Exclusion Criteria

1. There are signs of active infection/systemic illness going on, presence of fatigue and breathlessness even at rest.
2. Participant is febrile (body temperature >38.6degree Celsius)
3. Oxygen Saturation levels below <93%.
4. Systolic Blood pressure <90 mmHg or >180mmHg. -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Test | Baseline
  A simple 6 minutes' walk test (6MWT) is a reliable tool to assess cardiorespiratory effort tolerance in chronic lung and chronic heart failure patients. The test provides a global assessment of the cardio pulmonary reserves
6 Minutes Walk Test | 6th Week of Treatment
  A simple 6 minutes' walk test (6MWT) is a reliable tool to assess cardiorespiratory effort tolerance in chronic lung and chronic heart failure patients. The test provides a global assessment of the cardio pulmonary reserves
Rate of Perceived Exertion (RPE 6-20): | Baseline
  The Borg Rating of Perceived Exertion (RPE) scale is a subjective assessment of how hard someone feels they are working and can be helpful to guide people in choosing what activities to do as they progress through the phases of increasing physical activity.
Rate of Perceived Exertion (RPE 6-20): | 6th Week of Treatment
  The Borg Rating of Perceived Exertion (RPE) scale is a subjective assessment of how hard someone feels they are working and can be helpful to guide people in choosing what activities to do as they progress through the phases of increasing physical activity.
Post-Covid Functional Status Scale (PCFS) | Baseline
  An ordinal tool that is proposed to measure the full spectrum of functional outcomes following COVID-19
Post-Covid Functional Status Scale (PCFS) | 6th Week of Treatment
  An ordinal tool that is proposed to measure the full spectrum of functional outcomes following COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabiliation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelrahman Z, Li M, Wang X. Comparative Review of SARS-CoV-2, SARS-CoV, MERS-CoV, and Influenza A Respiratory Viruses. Front Immunol. 2020 Sep 11;11:552909. doi: 10.3389/fimmu.2020.552909. eCollection 2020. PMID 33013925
- [Background] Louis TJ, Qasem A, Abdelli LS, Naser SA. Extra-Pulmonary Complications in SARS-CoV-2 Infection: A Comprehensive Multi Organ-System Review. Microorganisms. 2022 Jan 12;10(1):153. doi: 10.3390/microorganisms10010153. PMID 35056603
- [Background] Siddiq MAB, Rathore FA, Clegg D, Rasker JJ. Pulmonary Rehabilitation in COVID-19 patients: A scoping review of current practice and its application during the pandemic. Turk J Phys Med Rehabil. 2020 Nov 9;66(4):480-494. doi: 10.5606/tftrd.2020.6889. eCollection 2020 Dec. PMID 33364571
- [Background] Calabrese M, Garofano M, Palumbo R, Di Pietro P, Izzo C, Damato A, Venturini E, Iesu S, Virtuoso N, Strianese A, Ciccarelli M, Galasso G, Vecchione C. Exercise Training and Cardiac Rehabilitation in COVID-19 Patients with Cardiovascular Complications: State of Art. Life (Basel). 2021 Mar 21;11(3):259. doi: 10.3390/life11030259. PMID 33801080
- [Background] Scudiero O, Lombardo B, Brancaccio M, Mennitti C, Cesaro A, Fimiani F, Gentile L, Moscarella E, Amodio F, Ranieri A, Gragnano F, Laneri S, Mazzaccara C, Di Micco P, Caiazza M, D'Alicandro G, Limongelli G, Calabro P, Pero R, Frisso G. Exercise, Immune System, Nutrition, Respiratory and Cardiovascular Diseases during COVID-19: A Complex Combination. Int J Environ Res Public Health. 2021 Jan 21;18(3):904. doi: 10.3390/ijerph18030904. PMID 33494244